CLINICAL TRIAL: NCT00581126
Title: Evaluation of Efficacy and Safety of Benefix®- Coagulation Factor ix, Recombinant, in Previously Treated Patients With Hemophilia b.
Brief Title: Study Evaluating BENEFIX in Previously Treated Patients With Hemophilia B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3090A-100932
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Hemophilia B
Keywords: BENEFIX; Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients will receive Benefix IV according to blood amount
  Interventions: Drug: Recombinant Factor IX Coagulation

INTERVENTIONS:
Drug: Recombinant Factor IX Coagulation — Benefix IV each 12 hours for 2 a 5 days

SUMMARY:
To assess efficacy and safety of BeneFix® for prophylaxis in "Short-term" therapy and on demand therapy for all bleeding episodes of subjects with hemophilia B.

DETAILED DESCRIPTION:
Phase IV, open-label, non comparative, multicenter, previously treated patients (PTP) clinical trial. Patients with severe or moderate hemophilia B with baseline levels of plasma factor IX < 5% activity will participate in this study for both treatment regimens: "on demand" therapy for acute bleeding episodes and therapy for prophylaxis of bleeding episodes ( "Short-term therapy")*.

* Short-Term Therapy: Prophylactic therapy given before surgery, including dental procedures, prior to a event that would likely result in bleeding ( sports, exercise, or heavy work), as well as to prevent further bleeds into a target joint). This short-term therapy for intermittent secondary therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with moderate to severe hemophilia B ( < 5% circulating factor IX activity) having acute hemorrhage or requiring "short-term therapy" for intermittent secondary prophylaxis regimens.
2. HIV seropositive ( asymptomatic) or seronegative subjects.
3. No history or detectable inhibitors.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2001-12; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
The primary variable will be the clinical response of BeneFix* in avoiding stopping or avoiding bleeding. | 9 months

SECONDARY OUTCOMES:
The secondary variables will be hemostasis and blood loss during and after surgery. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer